CLINICAL TRIAL: NCT01761357
Title: Impact of Burden of Comorbidities on Health Related Quality of Life Six Months After Transcatheter Aortic Valve Implantation in Patients Aged 75 Years and Older.
Brief Title: Burden Comorbidities and Transcatheter Aortic Valve Implantation
Acronym: TAVIQUAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RC12_0387
Record Dates: First submitted 2013-01-03; First posted 2013-01-04 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Symptomatic Severe Aortic Valve Stenosis in Older Patients
Keywords: Aortic valve stenosis; Quality of life; Burden co morbidities; Transcatheter aortic valve implantation; Geriatric assessment
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: answering to questionnaires of quality of live

SUMMARY:
The aim of the study is to determine whether the burden of comorbidities measured by CIRS-G (Cumulative Illness Rate Scale) is associated with a non-amelioration of the health related quality of life measured by questionnaire called "SF-36", six months after a transcatheter aortic valve replacement in older patients. During the comprehensive geriatric assessment realized before the valve implantation, the following data are recorded and their impact of the health related quality of life will also be analysed: comorbidity, age, depression, functional status, the cognitive impairment and malnutrition.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 75 years and older
* Patients referred for a transcatheter aortic valve implantation
* Patients who have a comprehensive geriatric assessment realized during the three months before the valve implantation
* Patients who provide informed written consent

Exclusion Criteria:

* Patients who refuse the study
* Patients with a legal guardian

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Difference of the physical component summary score of the health survey scale called "SF36", between inclusion and one month after the valve implantation. | 1 month

SECONDARY OUTCOMES:
Difference of the physical component summary score of the health survey scale called "SF36", between inclusion and three months after the valve implantation. | three months
Difference of the physical component summary score of the health survey scale called "SF36", between inclusion and six months after the valve implantation. | six months
Difference of the score of the Instrumental Activities of Daily Living scale called "IADL", between inclusion and one month after the valve implantation. | one month
Difference of the score of the Instrumental Activities of Daily Living scale called "IADL", between inclusion and three months after the valve implantation. | three months
Difference of the score of the Instrumental Activities of Daily Living scale called "IADL", between inclusion and six months after the valve implantation. | six months
Difference of the score of the Geriatric Depression Scale (GDS), between inclusion and one month after the valve implantation. | one month
Difference of the score of the Geriatric Depression Scale called "GDS", between inclusion and three months after the valve implantation | three months
Difference of the score of the Geriatric Depression Scale scale called "GDS", between inclusion and six months after the valve implantation | six months
Complications during the six months of follow up with all causes of mortality | 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Angers Universitary Hospital, Angers
  - Nantes Universitary Hospital, Nantes